CLINICAL TRIAL: NCT06067061
Title: "neoBREASTIM": A Phase 2 Study of Atezolizumab Plus RP1 Oncolytic Immunotherapy in the NeoAdjuvant Setting of Triple-Negative Breast Cancer (TNBC)
Brief Title: "neoBREASTIM": Atezolizumab Plus RP1 Oncolytic Immunotherapy in the NeoAdjuvant Setting of Triple-Negative Breast Cancer
Acronym: neoBREASTIM
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: Institut Curie (Other)
Collaborators: Replimune Inc. (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC 2021-10; 2022-502311-12-00 (Registry Identifier: EU trial number)
Record Dates: First submitted 2023-09-25; First posted 2023-10-04 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Triple Negative Breast Neoplasms
Keywords: Triple Negative Breast Cancer; Early-stage; Immunotherapy; Oncolytic virus
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — atezolizumab; MAPRE1 protein, human

STUDY DESIGN:
Intervention Model Description: An open-label, monocentric, single arm, phase II study with a safety run-in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab plus RP1 (Immulytic™) oncolytic immunotherapy (Experimental): Atezolizumab IV q2w RP1 (Immulytic™) by imaging-guided intra-tumor (IT) route.
  Interventions: Combination Product: Atezolizumab + RP1

INTERVENTIONS:
Combination Product: Atezolizumab + RP1 — Patients will be treated in a window period (ie 3 treatment cycles). After evaluation, patients that had no increase in ctDNA after 3 cycles (see Definition of ctDNA status) will continue on the same treatment (intratumoral injections of RP1 in combination with Atezolizumab) for a total of 10 treatment cycles prior to surgery.
  Other Names: Tecentriq®; Vusolimogene Oderparepvec

SUMMARY:
Neoadjuvant treatment is an important part of the treatment strategy for locally advanced TNBC having established a positive and significant correlation of pathologic Complete Response (pCR) with long-term clinical benefit such as Event-Free Survival (EFS) and Overall Survival (OS) as shown via large meta-analysis. Much effort has been made to identify novel agents and new drug combinations that can improve pCR rates in this specific clinical setting, which is the leading rationale to evaluate RP1 oncolytic immunotherapy in combination with Atezolizumab.

DETAILED DESCRIPTION:
The combination of RP1 plus Atezolizumab, while being expected to result in increased efficacy, is not expected to result in significant additional toxicity, as compared to either agent alone. Capitalizing on the strong prognostic and predictive value of the TIL infiltrate in early-stage TNBC and the capacity of circulating tumor DeoxyriboNucleic Acid (ctDNA) detection to predict response to immunotherapy and NeoAdjuvant Chemotherapy (NAC), neoBREASTIM - a single-arm phase 2 study - will evaluate a novel, biomarker-driven combination of Atezolizumab plus RP1 oncolytic immunotherapy in the neo-adjuvant setting of patients diagnosed with early-stage, TIL-high TNBC.

ELIGIBILITY:
Inclusion Criteria:

1. Female subject
2. Age ≥ 18 years old.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 1.
4. Newly diagnosed Triple-Negative Breast Cancer (TNBC), defined as the absence of estrogen expression and progesterone expression, and of Human Epidermal growth factor Receptor 2 (HER2) overexpression, must be determined by local testing of a screening tumor sample as defined by American Society of Clinical Oncology/College of American Pathologists guidelines.
5. TNBC defined as the following combined primary tumor (T), regional lymph node (N), and metastatic (M) American Joint Committee on Cancer staging criteria: cT ≥15 - ≤30 mm, N0, M0 according to Mammogram, breast Ultrasound and MRI, and PET-CT. In case of a difference in the measurement of the primary tumor among different imaging methods, the breast MRI measurement is the reference.
6. Unicentric, unifocal and unilateral disease.
7. Tumor-infiltrating lymphocytes (TILs) ≥ 30%, as defined by the International TILs Working Group 2014.
8. ctDNA dosing at baseline.
9. Agreement to provide tissue samples (tumor biopsy at screening and on-treatment), and at surgery for immune monitoring and translational research activities.
10. Agreement to perform blood samples at screening, on-treatment, and at surgery for immune monitoring and translational research activities.

Exclusion Criteria:

1. Inflammatory breast cancer.
2. Prior treatment with an oncolytic virus-based therapy.
3. Patients with active significant herpetic infections or prior complications of Herpes Simplex Virus-1 (HSV-1) infection.
4. Patients who require intermittent or chronic use of systemic (oral or IV) antivirals with known antiherpetic activity (e.g., acyclovir).
5. Diagnosis of immunodeficiency.
6. Has active autoimmune disease (e.g. inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, and multiple sclerosis, celiac disease, Wegener's granulomatosis) that has required systemic treatment in the past 3 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
7. Prior systemic immunosuppressive medication (except physiologic corticosteroid replacement therapy) within 30 days of planned start of study therapy.
8. Any live (attenuated) vaccine within 14 days of planned start of study therapy.
9. Prior immunotherapy, including tumor vaccine, cytokine, anti-CTLA4, PD-1/PD-L1 blockade or similar agents, T cell receptor-based (TCR-based) or Chimeric Antigen Receptor-T (CAR-T) cell based adoptive cell therapy.
10. Known history of, or any evidence of active, non-infectious pneumonitis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Safety of the combination Atezolizumab plus RP1 oncolytic during the safety run-in phase | 9 months
  Incidence of combination Atezolizumab plus RP1 adverse events (AEs) graded according to NCI CTCAE v5.0 and nature and severity
Toxicity of the combination Atezolizumab plus RP1 oncolytic immunotherapy during the safety run-in phase. | 9 months
  Dose Limiting Toxicity (DLT) during the first cycle of treatment of the combination Atezolizumab plus RP1 oncolytic immunotherapy
Residual Cancer Burden (RCB) 0-1 during the phase II part | 30 months
  Rate of RCB 0-1 at time of surgery (in patients with no increase in ctDNA after cycle 3)

SECONDARY OUTCOMES:
Response rate of RCB Score <= 1 at three cycles | 26 months
  Rate of RCB 0-1 after cycle 3 (in patients with no increase in ctDNA after cycle 3)
Safety and toxicity of the combination Atezolizumab plus RP1 oncolytic immunotherapy | 60 months
  Incidence, nature and severity of adverse events (AEs) graded according to NCI CTCAE v5.0 from the treatment start to the surgery
Invasive disease-free survival (iDFS) | 60 months
  iDFS will be measured using regular follow-up visits
Percentage of TILs | 30 months
  The percentage of TILs will be estimated and compared between RCB rates 0-1 versus 2-3
Pre-treatment expression of Programmed Death-Ligand 1 (PD-L1) | 30 months
  Expression of PD-L1 will be estimated and compared between RCB rates 0-1 versus 2-3
Correlation between RCB rates and response by Positron Emission Tomography-Scan (PET-CT) or breast MRI | 60 months
  To correlate the response by RCB rates with response by PET-CT or breast MRI will be studied
RCB rates and response | 60 months
  To correlate the response by breast MRI with RCB 0-1 rates,
Breast Conservation Surgery (BCS) | 30 months
  The rate of Breast Conservation Surgery (BCS) will be presented
Correlation between RCB rates and radiomics analyses | 30 months
  To correlate the RCB rates with response by radiomics analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Le Gouill, PhD, Study Director — Institut Curie
Locations (1):
- Institut Curie, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).